CLINICAL TRIAL: NCT04311437
Title: Effect of Self-acupressure on Middle Ear Barotrauma Associated With Hyperbaric Oxygen Therapy: a Nonrandomized Clinical Trial
Brief Title: Effect of Self-acupressure on Middle Ear Barotrauma Associated With Hyperbaric Oxygen Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: CMRPG8K0461
Record Dates: First submitted 2020-03-16; First posted 2020-03-17 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2021-07

CONDITIONS: Hyperbaric Oxygen Therapy; Middle Ear Barotrauma
Keywords: Hyperbaric oxygen therapy; Middle ear barotrauma; Acupressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-acupressure group (Experimental): The subjects in experimental group will undergo additional self-acupressure therapy in addition to Valsalva and Toynbee maneuvers before the first HBOT. The acupoints used are TE17 (Yifeng, 翳風), TE21 (Ermen, 耳門), SI19 (Tinggong, 聽宮), GB2 (Tinghui, 聽會).
  Interventions: Procedure: Self-acupressure therapy; Procedure: Combined Valsalva and Toynbee maneuvers
- Control group (Placebo Comparator): The subjects in control group will receive Valsalva and Toynbee maneuvers alone.
  Interventions: Procedure: Combined Valsalva and Toynbee maneuvers

INTERVENTIONS:
Procedure: Self-acupressure therapy — The self-acupressure therapy is as follows: Patients are in sitting position, applied firm pressure (3-5 kg of pressure) with the fingertips in a circular motion at a speed of two circles per second for a duration of one min per acupoint. A 1-2-s rest is applied after each ten circles. The complete process lasts for about 5 min.
  Arms: Self-acupressure group
Procedure: Combined Valsalva and Toynbee maneuvers — Valsalva maneuver: blowing against a closed mouth and nostrils, increasing the middle ear pressure. Toynbee maneuver: swallowing while the mouth and nostrils are closed, decreasing the middle ear pressure.

SUMMARY:
Middle ear barotrauma (MEB) is the most common complication during hyperbaric oxygen therapy (HBOT). Though Valsalva and Toynbee maneuvers have been proposed to prevent MEB, still some patients discontinue HBOT due to severe otalgia, hemorrhage or perforation of tympanic membrane associated with HBOT. Currently, there is no optimal prophylactic management for MEB associated with HBOT. The aim of this protocol is to investigate the efficacy of self-acupressure therapy on MEB associated with HBOT.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20 years or order receiving the first HBOT
* Alert consciousness

Exclusion Criteria:

* Pregnancy
* Having any acute disorder of the ears or upper respiratory tract
* Having evidence of neurologic dysfunction precluding them from making an informed decision
* Having a tracheostomy or endotracheal intubation
* Having received a myringotomy, tympanoplasty, mastoidectomy or tympanostomy tube placement.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Modified Teed Classification | 1 month
  The Modified Teed Classification, with grades from 0 to 5: Grade 0 indicates symptoms with no ontological signs of trauma; Grade 1 indicates injection of the tympanic membrane; Grade 2 indicates Grade 1 plus injection plus mild hemorrhage within the tympanic membrane; Grade 3 indicates gross hemorrhage within the tympanic membrane; Grade 4 indicates free blood in the middle ear as evidenced by blueness and bulging; and Grade 5 indicates perforation of the tympanic membrane.

SECONDARY OUTCOMES:
Symptoms of MEB | 1 month
  Record the symptoms of MEB including feeling pressure in the ears, ear pain, headache, dizziness, vertigo, tinnitus and hearing loss. Each symptom is estimated using a 10-cm visual analogue scale with anchor points of 0 (no discomfort) and 10 (maximum discomfort).
Overall ear discomfort levels | 1 month
  Estimated using a 10-cm visual analogue scale with anchor points of 0 (no discomfort) and 10 (maximum discomfort).

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Ting Liu, MD, Principal Investigator — Department of Chinese Medicine, Kaohsiung Chang Gung Memorial Hospital
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen JM, Lu ZN, Wu RW, Bi KW, Liu CT. Effect of self-acupressure on middle ear barotrauma associated with hyperbaric oxygen therapy: A nonrandomized clinical trial. Medicine (Baltimore). 2021 Apr 30;100(17):e25674. doi: 10.1097/MD.0000000000025674. PMID 33907136